CLINICAL TRIAL: NCT05057546
Title: Ovarian Hormone Regulation of Central and Cerebrovascular Hemodynamics
Brief Title: Ovarian Hormone Regulation of Central and Cerebrovascular Hemodynamics (NoMEN Study)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-3590
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Menopause; Estrogen Deficiency; Women; Aging
MeSH Terms: interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Intervention Model Description: BESH clinical trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Premenopausal Group: GnRH antagonist (Experimental): Gonadotropin releasing hormone (GnRH) antagonist is degarelix acetate, 80 mg, delivered once as a subcutaneous injection.
  Interventions: Drug: GnRH antagonist

INTERVENTIONS:
Drug: GnRH antagonist — GnRH antagonist will be given once for premenopausal women (12-week intervention) and twice for postmenopausal women (24-week intervention)
  Other Names: Degarelix acetate

SUMMARY:
This study will evaluate changes in blood vessels around the heart (e.g., aorta and carotid arteries) and in the brain with the loss of female sex hormones (e.g., estrogen) during the menopause transition. The menopause transition is associated with declines in blood vessel function and increased risk for cardiovascular disease and Alzheimer's disease. Increasing evidence supports an early role for declines in blood vessel function and future development of Alzheimer's disease in aging men and women. This study will learn about the effects of changes in female sex hormones, such as estrogen, during the menopause transition on blood vessel around the heart and in the brain in women.

ELIGIBILITY:
Inclusion Criteria: Healthy premenopausal, early perimenopausal and postmenopausal women will be recruited. Premenopausal women will have regular menstrual cycles, with no change in observed cycle length (21-35 days), confirmed by menstrual cycle calendars. Early perimenopausal will be defined as a change in cycle length of >7 days from normal with no skipped periods and/or a FSH <25 IU/L (with discretion of the study MD). Postmenopausal women will have gone through natural (i.e., non-surgical) menopause with >12 months but <6 years of amenorrhea. We will make a major effort to ensure that the women enrolled in this study come from all races and ethnicities and a wide range of socioeconomic and educational levels.

Exclusion Criteria:

* Seated resting blood pressure >140/90 mmHg
* Use of medications that might influence cardiovascular function or cerebral blood flow;
* Pregnant, currently breastfeeding or intention to become pregnant in the next 6 months;
* Use of menopausal therapy or hormonal contraceptives, etc. within the previous 3 months or intent to start during the study period;
* BMI >39 kg/m2;
* Vigorous intensity exercise >2 days per week;
* Any current or past history of systemic illness that would interfere with study outcomes such as: diabetes, cancer (other than melanoma), liver, gallbladder disease, peripheral artery disease or thromboembolism, neurological disease, CVD or cerebrovascular disease;
* Abnormal thyroid, liver, or kidney function testing during the screening examination or bloodwork;
* Plasma glucose >126 mg/dl under fasting conditions;
* Smoking or living with a smoker within the past 12 months;
* Current or planned participation in an interventional study during the present study or unwillingness to complete study-related procedures;
* Patients who report active acute systemic infection (e.g., flu, common cold, etc), fever (> 100.0 °F) or feeling ill will be asked to delay vascular testing until they are no longer febrile or ill. Additionally, anyone who has experienced a serious illness (requiring hospitalization) within the last 6 months, had a confirmed positive COVID test and hospitalized, or anyone with a confirmed positive COVID test within the last 6 months will be ineligible to participate (discretion of the study PI and MD).
* No use of vitamin/supplements or chronic use of anti-inflammatory medications, or willingness to stop 1 month prior to the vascular visit.

In premenopausal women participating in the intervention:

* Contraindications to Degarelix including hypersensitivity to degarelix acetate, extrinsic peptide hormones, mannitol, GnRH, benzyl alcohol (the vehicle for injection of degarelix acetate)
* Undiagnosed vaginal bleeding
* Osteopenia or osteoporosis (i.e., proximal femur or lumbar spine DXA Z scores <-1.0)
* CES-D score ≥16 (unless clinician follow-up and clinical judgement determine they are eligible (will be noted in study chart)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2025-07-28 (Estimated)

PRIMARY OUTCOMES:
Aortic stiffness and pulsatile hemodynamics | Change from baseline at 12 weeks
  Aortic characteristic impedance and forward pressure wave amplitude

SECONDARY OUTCOMES:
Common carotid artery stiffness and pulsatile hemodynamics | Change from baseline at 12 weeks
  Carotid characteristic impedance and forward pressure wave amplitude
Macrovascular cerebral blood flow | Change from baseline at 12 weeks
  Cerebral blood flow measured by transcranial Doppler
Macrovascular cerebrovascular reserve | Change from baseline at 12 weeks
  Breath hold index measured by transcranial Doppler
Microvascular cerebral blood flow | Change from baseline at 12 weeks
  Cerebral blood flow measured by Arterial Spin Labeling Magnetic Resonance Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Lyndsey DuBose, PhD, Principal Investigator — University of Colorado Denver Anschutz Medical Campus
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No